CLINICAL TRIAL: NCT03916510
Title: A Phase 1 Trial of the Safety, Tolerability and Biological Effects of Intravenous Enadenotucirev, a Novel Oncolytic Virus, in Combination With Chemoradiotherapy in Locally Advanced Rectal Cancer
Brief Title: Chemoradiation With Enadenotucirev as a Radiosensitiser in Locally Advanced Rectal Cancer
Acronym: CEDAR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Akamis Bio (Industry); Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OCTO_081
Record Dates: First submitted 2019-04-09; First posted 2019-04-16 (Actual); Results first posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2023-04

CONDITIONS: Locally Advanced Rectal Cancer
Keywords: locally advanced; rectal cancer; Enadenotucirev; oncolytic virus; adenovirus; dose escalation; Time To Event Continual Reassessment Method; chemoradiotherapy; phase 1
MeSH Terms: conditions — Rectal Neoplasms; Adenoviridae Infections | interventions — enadenotucirev; Capecitabine; Radiotherapy

STUDY DESIGN:
Intervention Model Description: CEDAR is a dual escalation phase 1 trial using a TiTE CRM (Time To Event Continual Reassessment Method).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dosing Group 1 (Experimental): * Chemotherapy: 900 mg/m2 capecitabine twice daily, Mon-Fri (on radiotherapy days) for 5 weeks, except on days patients received enadenotucirev.
  * Radiotherapy: 50 Gy in 25 fractions.
  * Enadenotucirev: 3 x loading doses pre-chemoradiation (low-low-low*).
    * Low = 1x10^12 viral particles High = 3x10^12 viral particles
  Interventions: Biological: Enadenotucirev; Drug: Capecitabine; Radiation: Radiotherapy
- Dosing Group 2 (Experimental): * Chemotherapy: 900 mg/m2 capecitabine twice daily, Mon-Fri (on radiotherapy days) for 5 weeks, except on days patients received enadenotucirev.
  * Radiotherapy: 50 Gy in 25 fractions.
  * Enadenotucirev: 3 x loading doses pre-chemoradiation (low-low-low*). 3 x maintenance doses post-chemoradiation (low-low-low*).
    * Low = 1x10^12 viral particles High = 3x10^12 viral particles
  Interventions: Biological: Enadenotucirev; Drug: Capecitabine; Radiation: Radiotherapy
- Dosing Group 3 (Experimental): * Chemotherapy: 900 mg/m2 capecitabine twice daily, Mon-Fri (on radiotherapy days) for 5 weeks, except on days patients received enadenotucirev.
  * Radiotherapy: 50 Gy in 25 fractions.
  * Enadenotucirev: 3 x loading doses pre-chemoradiation (low-low-low*). 3 x maintenance doses post-chemoradiation (low-high-high*).
    * Low = 1x10^12 viral particles High = 3x10^12 viral particles
  Interventions: Biological: Enadenotucirev; Drug: Capecitabine; Radiation: Radiotherapy
- Dosing Group 4 (Experimental): * Chemotherapy: 900 mg/m2 capecitabine twice daily, Mon-Fri (on radiotherapy days) for 5 weeks, except on days patients received enadenotucirev.
  * Radiotherapy: 50 Gy in 25 fractions.
  * Enadenotucirev: 3 x loading doses pre-chemoradiation (low-high-high*). 2 x concurrent doses on week 1, days 1 and 5 of chemoradiation (high-high*). 3 x maintenance doses post-chemoradiation (low-high-high*).
    * Low = 1x10^12 viral particles High = 3x10^12 viral particles
  Interventions: Biological: Enadenotucirev; Drug: Capecitabine; Radiation: Radiotherapy

INTERVENTIONS:
Biological: Enadenotucirev — Enadenotucirev is a live replicating oncolytic adenovirus; it is considered a BioSafety Level 1 (BSL-1) infectious substance.
Drug: Capecitabine — Capecitabine is a chemotherapy drug licensed for use in rectal cancer, it is a non-cytotoxic pre-cursor of the cytotoxic 5-fluorouracil. Due to Capecitabine not being taken on Enadenotucirev dosing days it is considered an investigational medicinal product within this trial.
Radiation: Radiotherapy — 50 Gy/25#

SUMMARY:
The use of chemoradiotherapy (CRT), in combination with surgery is the standard of care in the treatment of locally advanced rectal cancer. However some patients don't respond well to radiation.

More advanced radiotherapy techniques, that result in fewer toxicities, means that we are now able to combine new anti-cancer agents into standard treatment. Targeting the tumour early in this way has the potential to improve response rates.

Enadenotucirev is a specific type of anti-cancer virus that only targets cancer cells. It acts in the same way as any virus and can only survive by replicating inside cancer cells and not normal, non-cancerous cells. This means that it can selectively target and destroy tumours, without directly affecting normal cells. It also has the ability to attract cells from the body's immune system to help fight the cancer.

The addition of enadenotucirev to standard chemoradiotherapy treatment may have a combined effect on the cancer cells with potentially few, additional side effects.

This trial aims to determine the optimal dose and frequency of the virus to give by gradually increasing the number of doses each successive patient receives, and then increasing the dose of the virus itself. Each patient will receive a minimum of 3 doses, up to a maximum of 8, spread over the course of their 5 week standard chemoradiotherapy treatment. Patients will be closely monitored at all times to ensure that with each dosing group, there aren't excessive side effects.

Patients will then undergo surgery as part of their standard of care and be followed up for up to 4-6 weeks post-surgery.

This trial aims to determine the optimal dose and frequency that can then be used in future studies with the possibility of exploring the addition of Enadenotucirev to other chemoradiotherapy treatments.

DETAILED DESCRIPTION:
At present identifying novel radiosensitising agents in colorectal cancer is an area of high need for patients considering sphincter preserving surgery or needing down staging to facilitate surgery.

Although the combination of Enadenotucirev with chemoradiation is novel, there is a wealth of evidence to support the rationale for combining this class of agent with radiation and chemotherapy.

Enadenotucirev is a group B oncolytic virus under development for the systemic treatment of metastatic or advanced epithelial tumours. Enadenotucirev is a chimeric adenovirus type 11p (Adp/adenovirus type 3 (Ad3) virus, discovered through a process of bio-selection from a library of chimeric viruses produced from a pool of adenoviruses from seven different serotypes utilizing human HT-29 colorectal cancer (CRC) cells.

Enadenotucirev shows selective and potent toxicity in humans carcinoma cells with only very limited or no toxicity to normal (non-cancerous) human cells. Other than humans, there is no known permissive species for Enadenotucirev. The principle advantage of oncolytic therapy is that the virus replicates only in diseased cells meaning that the concentration of drug is amplified at the site of pathology so that it is higher in the tumour than in healthy tissue. Virus particles spread from cell to cell within a tumour nodule until they reach non-permissive normal tissues, in principle destroying all viable tumour cells they encounter.

While the overall understanding of the mechanism of action of Enadenotucirev in humans is still under investigation, it is now well established from non-clinical and clinical studies that the mechanism of anti-cancer efficacy of oncolytic viruses not only involves direct infection and lysis of tumour cells, but that immune responses stimulated via an increased release of tumour-associated antigens and immune-inflammatory activation signals play a key role.

CEDAR is dual endpoint, dose escalation phase 1 trial using a time to event continual reassessment method (TiTE CRM). Response and Toxicity endpoints will be combined in dose escalation models to identify the optimal dose schedule. Dose decisions are made using the statistical model which uses number of Dose Limiting Toxicities (DLT) experienced in different dosing schedules, instead of just using the data from that particular dose, as in the case of 3+3 model, meaning it uses all available data to make a dose decision.

This primary objective is to determine the optimal dose and frequency of the virus by firstly gradually increasing the number of doses each successive patient receives, and then increasing the dose of the virus itself. All participants will receive 3 loading doses in weeks 1-2, prior to initiation of standard chemoradiotherapy. Further doses of Enadenotucirev will either be given after or during and after standard chemoradiotherapy and this is dependent on which of the 4 different dose groups they are assigned to. The individual doses given will be either 1x10^12 viral particles (vp) or 3x10^12 vp.

Each patient will receive a minimum of 3 doses, up to a maximum of 8, spread over the course of 9 weeks. Patients will be closely monitored at all times to ensure that with each dosing group, there aren't excessive side effects.

Patients will then undergo surgery as part of their standard of care and be followed up for 4-6 weeks after surgery.

Dose Limiting Toxicities (DLTs)

DLTs are defined as any of the following occurring between the start of trial treatment until the Week 13 visit and assessed as possibly, probably or definitely related to enadenotucirev or the interaction between enadenotucirev and radiotherapy and/or capecitabine.

Renal:

o Development of proteinuria, 2+ as measured by urinalysis and confirmed with an albumin/creatinine ratio of >3g/mmol with a 24-hour urinary protein ≥1g/24h or if there is a decline in estimated glomerular filtration rate (eGFR) (where a decline in eGFR is defined as eGFR <60ml/min/1.73m2 or a drop in eGFR by 20% from screening, baseline of previous visit), following administration of enadenotucirev, shall be classified as a DLT. No further doses of enadenotucirev will be administered to that patient.

Acute hematologic toxicity:

* Infection (documented clinically or microbiologically) with grade 3 or 4 neutropenia (absolute neutrophil count (ANC) <1.0 x 10^9/L)
* Neutropenia grade 4 (ANC < 0.5 x 10^9/L) lasting for ≥7 days
* Febrile neutropenia grade 4 (fever of unknown origin without clinically or microbiologically documented infection) (ANC <1000/mm3 with a single temperature of >38.3 degrees Celsius or a sustained temperature of >=38 degrees Celsius for more than one hour)
* Thrombocytopenia grade 3 (Platelet count < 50 x 10^9/L) in the presence of bleeding or requiring platelet transfusion
* Thrombocytopenia grade ≥ 4 (Platelet count < 25 x 10^9/L)
* Anemia grade 3 in the presence of blood transfusion dependency as judged by the Principal Investigator
* Anemia grade ≥ 4
* Clinically significant bleeding attributed to grade 3 thrombocytopenia or requiring platelet transfusion or other grade ≥3 clotting disorder or occurring concurrently with Grade 2 or 3 activated partial thromboplastin time (aPTT) prolongation, unless there is a clear explanation for the event, such as tumour-related bleeding in the presence of Lupus Anticoagulant.
* Any other grade ≥3 non-hematological toxicity with the exception of: aPTT prolongation
* Clotting event (i.e. deep vein thrombosis, pulmonary embolism) occurring concurrently with Grade 2 or 3 aPTT prolongation

Acute non-hematologic toxicity:

* Any documented ≥ grade 4 non-hematologic toxicity in the presence of maximal support/active management
* Grade ≥3 cystitis or radiation dermatitis onset within 2 weeks of starting radiotherapy or lasting more than 2 weeks after the end of radiotherapy
* Grade ≥3 proctitis or diarrhea onset within 2 weeks of starting radiotherapy
* Grade ≥3 nausea or vomiting not controlled by optimal outpatient anti-emetic treatment
* Grade ≥3 diarrhea despite optimal outpatient anti-diarrheal medication use
* Grade ≥3 hematuria or neuropathic pain
* Other grade 3 ≥ effects thought to be due to the combination of enadenotucirev with radiotherapy
* Missing 2 consecutive doses of enadenotucirev due to enadenotucirev toxicity
* An elevation of alanine transaminase (ALT) or aspartate aminotransferase (AST) >5 x upper limit of normal lasting 8 days or more
* A concurrent elevation of ALT or AST >3 × upper limit of normal and total bilirubin >2 × upper limit of normal in whom there is no evidence of biliary obstruction or other causes that can reasonably explain the concurrent elevation
* Death due to drug related complications
* Grade ≥3 cytokine release syndrome

General:

* Discontinuation of the active treatment due to toxicity definitely attributable to enadenotucirev, irrespective of the grade of toxicity
* Missing 3 consecutive fractions of radiotherapy, related to enadenotucirev, as judged by the Principal Investigator
* Any toxicity causing a delay of radiotherapy completion by greater than one week

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed invasive adenocarcinoma of the rectum
2. Locally advance colorectal cancer as defined by pelvic MRI with a threatened circumferential resection margin (cT3mrf+ve), or inclusion of an adjacent organ, or low tumours at/below the level of the levators or enlarged pelvic side wall nodes or selected by the multidisciplinary team MDT for treatment with neoadjuvant (chemo)radiotherapy, regardless of TNM classification
3. Patients with oligometastatic disease suitable for radical treatment are permitted provided that the site specific MDT deems them suitable for chemoradiation
4. Male or female, Age ≥ 18 years
5. ECOG performance score of 0 - 1
6. The patient is willing and able to comply with the protocol scheduled biopsy, follow-up visits and examinations for the duration of the trial.
7. Written (signed and dated) informed consent
8. Adequate renal function demonstrated by:

   * Adequate ≤1.5 ULN and estimated glomerular filtration rate (eGFR) ≥60 mL/min/1.73m (measured creatinine clearance ≥60 mL/min) and
   * Urine dipstick for proteinuria at screening and baseline negative or trace. Patients may be included with results of 1+ if they have a spot urinary albumin creatinine ratio (ACR) of either:

     (i) ≤3 mg/mmol or (ii) >3 mg/mmol with a 24 hour urinary protein <1.0 g/24 hours and
   * Serum complement C3 and C4 within the normal range
9. Haematological and Biochemical indices within the ranges shown below:

   * Haemoglobin: ≥90 g/L
   * Absolute neutrophil count: ≥1.5x10^9/L
   * Platelet count: ≥100x10^9/L
   * Bilirubin: < 1.5 upper limit of normal
   * Aspartate transaminase and/or alanine transaminase: ≤3 x upper limit of normal
   * INR: ≤1.5
   * aPTT: within laboratory normal range

Exclusion Criteria:

1. Pregnant or breast-feeding women, or women of childbearing potential unless effective methods of contraception are used.
2. Pulmonary lymphangitis (if metastatic disease present)
3. Past medical history:

   1. Known history or evidence of significant immunodeficiency due to underlying illness and/or medication (e.g. systemic corticosteroids, or other immunosuppressive medications including cyclosporine, azathioprine, interferons in the 4 weeks before the first dose of trial treatment)
   2. Splenectomy
   3. Prior allogeneic or autologous bone marrow or organ transplantation
   4. Patients with a history of, or active, known or suspected auto-immune disease or a syndrome that requires systemic or immunosuppressive agents; patients with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune disease only requiring hormone replacement, psoriasis not requiring systemic treatment or conditions not expected to recur in the absence of an external trigger are permitted to enrol.
   5. History of idiopathic pulmonary fibrosis, drug-induced pneumonitis, or evidence of active pneumonia or pneumonitis on computed tomography scan
   6. Active viral disease or known positive serology for HIV, hepatitis B or hepatitis C
   7. Active infections requiring antibiotics, physician monitoring, or recurrent fevers >38.0°C associated with a clinical diagnosis of active infection
   8. Prior pelvic radiotherapy
   9. Any other active malignancy, with the exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri and non-melanoma skin lesions
   10. Uncontrolled cardiorespiratory comorbidity (e.g. severe pulmonary fibrosis, inadequately controlled angina or myocardial infarction in the last 6 months)
   11. Major disturbance in bowel function (e.g. severe incontinence, Crohn's disease, >6 loperamide/day), risk of bowel obstruction due to tumour - exception defunctioning colostomy performed
   12. Treatment with any COVID-19 vaccine in the 28 days before the first dose of enadenotucirev, unless the vaccine is known to not be based on an adenoviral vector (e.g. mRNA vaccines)
   13. Treatment with any vaccine (including known non-adenoviral COVID-19 vaccines) in the 7 days before first dose of enadenotucirev
4. Use of the following anti-viral agents: ribavirin, adefovir, lamivudine or cidofovir within 7 days prior to the first dose of trial treatment
5. Treatment with any other investigational agent, or participation in another interventional clinical trial within 28 days prior to enrolment. In follow up for an interventional trials and observational studies are allowed
6. History of DVT or pulmonary embolus in the 12 months before the first dose of study of study treatment
7. History of significant bleeding requiring hospitalisation in the 12 months before the first dose of study treatment
8. Patients receiving therapeutic or prophylactic anticoagulation therapy
9. Known dihydropyrimidine dehydrogenase (DPYD) deficiency
10. Prior chemotherapy is allowed as long as >28 days since the last administration and any toxicity has resolved to NCI CTCAE grade 1 or less
11. Other psychological, social or medical condition, physical examination finding or a laboratory abnormality that the investigator considers would make the patient a poor trial candidate or could interfere with protocol compliance or the interpretation of trials results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Hawkins, MD FRCR MRCP, Principal Investigator — University of Oxford
Locations (4):
- United Kingdom (4):
  - Velindre Cancer Centre, Cardiff
  - Beatson West Of Scotland Cancer Centre, Glasgow
  - The Churchill Hospital, Oxford University Hospitals Trust, Oxford
  - Royal Marsden NHS Foundation Trust, Sutton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] O'Cathail SM, Davis S, Holmes J, Brown R, Fisher K, Seymour L, Adams R, Good J, Sebag-Montefiore D, Maughan T, Hawkins MA. A phase 1 trial of the safety, tolerability and biological effects of intravenous Enadenotucirev, a novel oncolytic virus, in combination with chemoradiotherapy in locally advanced rectal cancer (CEDAR). Radiat Oncol. 2020 Jun 12;15(1):151. doi: 10.1186/s13014-020-01593-5. PMID 32532291

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was registered on 29Jul2019 and the final study visit for the final patient was on 28Oct2022.
Groups:
- Dosing Group 3: * Chemotherapy: 900 mg/m2 capecitabine twice daily, Mon-Fri (on radiotherapy days) for 5 weeks, except on days patients received enadenotucirev.
  * Radiotherapy: 50 Gy in 25 fractions.
  * Enadenotucirev: 3 x loading doses pre-chemoradiation (low-low-low)*. 3 x maintenance doses post-chemoradiation (low-high-high)*.
    * Low = 1x10^12 viral particles High = 3x10^12 viral particles
Period: Overall Study
Arm/Group | Dosing Group 1 | Dosing Group 2 | Dosing Group 3 | Dosing Group 4
Started | 2 | 4 | 6 | 0
Completed | 2 | 4 | 6 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Dosing group 4 was a planned schedule of treatment per protocol. However, the data collected during the trial, did not warrant escalation to this schedule, therefore there were no participants registered to this dosing group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dosing Group 1 | Dosing Group 2 | Dosing Group 3 | Dosing Group 4 | Total
Number analyzed (Participants) | 2 | 4 | 6 | 0 | 12
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 42.0 [36.5 to 47.5] | 65.5 [59.0 to 68.2] | 63.5 [54.0 to 72.2] |  | 61.0 [50.5 to 70.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 |  | 3
  Male | 1 | 3 | 5 |  | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
ECOG Performance Status [Count of Participants; unit: Participants] — ECOG (Eastern Cooperative Oncology Group) Performance Status assesses the functional status of a patient (ref: Oken MM, et al. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-655).
  All participants in the trial were assessed as ECOG status 0 or 1.
  0 = Fully active, able to carry on all pre-disease performance without restriction
  1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  Participants
    ECOG performance status = 0 | 2 | 4 | 5 |  | 11
    ECOG performance status = 1 | 0 | 0 | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had a Dose Limiting Toxicity (DLT) Following Treatment With Enadenotucirev and Chemoradiotherapy (Capecitabine and Radiation) at 1 of 4 Different Dosing Schedules.
Description: Dose escalation for this trial was informed by a Time To Event Continual Reassessment Method (TiTE CRM). This statistical model was also able to determine the optimal dose schedule of enadenotucirev that can be administered with chemoradiation (highest treatment schedule resulting in less than 30% dose limiting toxicity rate). The definition of a DLT for this trial can be found in the study description section of this record.
Time Frame: From Day 1 of treatment to Week 13 (13 weeks +/- 3 days)
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Dosing Group 1 | Dosing Group 2 | Dosing Group 3 | Dosing Group 4
Number analyzed (Participants) | 2 | 4 | 6 | 0
participants | 0 | 0 | 1 |

2. Primary Outcome: Magnetic Resonance Imaging (MRI) Tumour Regression Grade on a Scale of 1-5 for Patients Treated With Enadenotucirev Delivered in Conjunction With Chemoradiotherapy (Capecitabine and Radiation) at 1 of 4 Different Dosing Schedules.
Description: To inform the optimal dose and frequency of enadenotucirev that can be administered with chemoradiation. The MRI tumour regression grade uses the following scale and for the purposes of the trial analysis and dose escalation, scores of 1 or 2 were classified as responders and scores of 3, 4 or 5 were classified as non-responders:
  1. - No/minimal fibrosis visible (tiny linear scar) and no tumour signal (best outcome)
  2. - Dense fibrotic scar (low signal intensity) but no macroscopic tumour signal (indicates no or microscopic tumour)
  3. - Fibrosis predominates but obvious measurable areas of tumour signal visible
  4. - Tumour signal predominates with little/minimal fibrosis
  5. - Tumour signal only: no fibrosis, includes progression of tumour (worst outcome)
Time Frame: 13 weeks after starting treatment (+/- 3 days)
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Dosing Group 1 | Dosing Group 2 | Dosing Group 3 | Dosing Group 4
Number analyzed (Participants) | 2 | 4 | 6 | 0
participants
  1 - No/minimal fibrosis visible (tiny linear scar) and no tumour signal (best outcome) | 0 | 0 | 1 |
  2 - Dense fibrotic scar but no macroscopic tumour signal (indicates no or microscopic tumour) | 0 | 2 | 2 |
  3 - Fibrosis predominates but obvious measurable areas of tumour signal visible | 0 | 1 | 3 |
  4 - Tumour signal predominates with little/minimal fibrosis | 2 | 1 | 0 |
  5 - Tumour signal only: no fibrosis, includes progression of tumour (worst outcome) | 0 | 0 | 0 |

3. Secondary Outcome: Number of Patients Completing at Least 80% of the Intended Capecitabine Dose and at Least 20 Fractions of Radiotherapy.
Description: Ability to deliver enadenotucirev concurrently with chemoradiation, based on treatment tolerance for the combination of enadenotucirev, capecitabine and radiation.
Time Frame: From start of treatment to end of treatment (9 weeks)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Dosing Group 1 | Dosing Group 2 | Dosing Group 3 | Dosing Group 4
Number analyzed (Participants) | 2 | 4 | 6 | 0
Participants
  Received > 80% of intended capecitabine dose and at least 20 fractions of radiotherapy | 2 | 4 | 5 |
  Did not receive > 80% of intended capecitabine dose and at least 20 fractions of radiotherapy | 0 | 0 | 1 |

4. Secondary Outcome: Number of Participants With Pathological Complete Response (pCR) of Tumour Following Resection (Staged According to Royal College of Pathologists Guidelines).
Description: To measure local response rate to combined therapy following treatment with enadenotucirev, capecitabine and radiotherapy. Pathological complete response (pCR) was only observable in patients undergoing surgery. The final resected tumour was assessed by an experienced lower gastrointestinal pathologist and staged according to the Royal College of Pathologists recommended standard datasets as per standard of care. Pathological complete response (pCR) is staged as ypT0N0 - a complete regression of the primary tumour (ypT0), with concurrently no (residual) tumoral invasion of the lymph nodes (ypN0).This notation is part of the TNM staging system used in oncology, where "T" stands for the size and extent of the main tumour, and "N" describes the presence of cancer in nearby lymph nodes.
Time Frame: At 4-6 weeks post surgery (minimum 18 weeks after start of treatment)
Population: Dosing group 4 was a planned schedule of treatment per protocol. However, the data collected during the trial, did not warrant escalation to this schedule, therefore there were no participants registered to this dosing group. In addition, there were 2 participants in dosing group 2 and 2 participants in dosing group 3 who did not have surgery, and therefore were not included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Dosing Group 1 | Dosing Group 2 | Dosing Group 3 | Dosing Group 4
Number analyzed (Participants) | 2 | 2 | 4 | 0
Participants
  Pathological complete response = yes | 0 | 0 | 1 |
  Pathological complete response = no | 2 | 2 | 3 |

5. Secondary Outcome: Neoadjuvant Rectal (NAR) Score on a Scale of 0-100 Following Resection.
Description: To measure local response rate to combined therapy following treatment with enadenotucirev, capecitabine and radiotherapy. The Neoadjuvant Rectal (NAR) score ranges from 0-100, where a higher score equates to a worse prognosis. The NAR score outperforms pathological complete response (pCR) at predicting disease free survival (DFS) and overall survival (OS) in clinical trials using neoadjuvant therapy for rectal cancer. It similarly performs well at predicting DFS and OS in trials using pre-op chemo and chemoradiotherapy. Ref: George TJ, Allegra CJ, Yothers G. Neoadjuvant Rectal (NAR) Score: a New Surrogate Endpoint in Rectal Cancer Clinical Trials. Curr Colorectal Cancer Rep. 2015;11(5):275-80.
  NAR = [5pN - 3(cT - pT) + 12]^2 / 9.61
  Where:
  cT is an element of the set {1, 2, 3, 4}, pT is in {0, 1, 2, 3, 4}, pN is in {0, 1, 2}. cT clinical tumour stage, pT pathologic tumour stage, pN pathologic nodal stage
Time Frame: At 4-6 weeks post surgery (minimum 18 weeks after start of treatment)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Neoadjuvant Rectal (NAR) score
Arm/Group | Dosing Group 1 | Dosing Group 2 | Dosing Group 3 | Dosing Group 4
Number analyzed (Participants) | 2 | 2 | 4 | 0
Neoadjuvant Rectal (NAR) score | 22.5 (10.7) | 15.0 (0.0) | 17.0 (22.5) |

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from the time patients consented to the trial until they completed their 4-6 weeks post-surgery visit (minimum duration 18 weeks).
Description: Dosing group 4 was a planned schedule of treatment per protocol. However, the data collected during the trial, did not warrant escalation to this schedule, therefore there were no participants registered to this dosing group and thus, no patients were at risk in this group and adverse events were collected.
Arm/Group | Dosing Group 1 | Dosing Group 2 | Dosing Group 3 | Dosing Group 4
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/4 | 1/6 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/4 | 2/6 | 0/0
Other Adverse Events (participants affected / at risk) | 2/2 | 4/4 | 6/6 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dosing Group 1 (N=2) | Dosing Group 2 (N=4) | Dosing Group 3 (N=6) | Dosing Group 4 (N=0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dosing Group 1 (N=2) | Dosing Group 2 (N=4) | Dosing Group 3 (N=6) | Dosing Group 4 (N=0)
Neutropenia (Blood and lymphatic system disorders) | 1 (4) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Radiation skin injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Balanoposthitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Anal pruritus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anorectal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (4) | 3 (6) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Faeces soft (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Rectal tenesmus (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 2 (4) | 5 (9) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 5 (5) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cystitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Polydipsia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (General disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tension (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysparaeunia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral coldness (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-05-05): https://cdn.clinicaltrials.gov/large-docs/10/NCT03916510/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-04): https://cdn.clinicaltrials.gov/large-docs/10/NCT03916510/SAP_001.pdf